CLINICAL TRIAL: NCT02485054
Title: Development and Validation of a Predictive Score for the Ischemic Etiology of a Transient Visual Disturbances
Brief Title: A Predictive Score for the Ischemic Etiology of a Transient Visual Disturbances (VASCO)
Acronym: VASCO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MOA_2014-32
Record Dates: First submitted 2015-06-18; First posted 2015-06-30 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Eligible patients: Adults having had a transient visual disturbance during the last 8 days, except a diplopia
  Interventions: Other: Clinical, ophthalmological and neurological evaluation

INTERVENTIONS:
Other: Clinical, ophthalmological and neurological evaluation — Clinical : questionnaire about the symptoms and about the vascular risk factors Cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography

SUMMARY:
The transient visual disturbances (TVD) are defined by a short abnormality of visual function. Their etiology may be ophthalmological, neurological non-ischemic or of ischemic origin.

The difficulty is to recognize an ischemic mechanism which imposes emergency cares.

A clinical score could help the clinician to recognize the etiology of the TVD .

ELIGIBILITY:
Inclusion Criteria:

* Transient visual disturbances (i.e. less than 24 hours) during the last 8 days

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults having had a transient visual disturbance during the last 8 days and seen at the fondation ophtalmologique Adolphe de Rothschild
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Etiology, ischemic or not, of the initial transient visual disturbance | 3 months
  Clinical : questionnaire about the symptoms and about the vascular risk factors Cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.

SECONDARY OUTCOMES:
Incidence of new visual transient ischemic attacks during the 3 months of follow-up | 3 months
  Clinical : questionnaire about the symptoms and about the vascular risk factors Cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.
Incidence of visual ischemic strokes during the 3 months of follow-up | 3 months
  Clinical : questionnaire about the symptoms and about the vascular risk factors Cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.
Incidence of transient ischemic attacks, visual or not visual, during the 3 months of follow-up | 3 months
  Clinical : questionnaire about the symptoms and about the vascular risk factors Cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.
Incidence of ischemic strokes, visual or not visual, during the 3 months of follow-up | 3 months
  Clinical : questionnaire about the symptoms and about the vascular risk factors Cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Bichat, Paris
  - Fondation ophtalmologique Adolphe de Rothschild, Paris